CLINICAL TRIAL: NCT05552066
Title: Before and After Study, Evaluating the Efficiency of an Anticipated Personalization of the Management in Day Hospital Unit Based on a Collection of the PROs Via a Digital Tool
Brief Title: Anticipated Personalization of the Management in Day Hospital Unit Based on a Collection of the PROs Via a Digital Tool
Acronym: ANTICIPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-3-29-001
Record Dates: First submitted 2022-09-07; First posted 2022-09-23 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Solid Malignant Tumor
Keywords: PRO (Patient reported outcomes); Chemotherapy; immunotherapy; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: 1st stage: the current circuit remains unchanged (with sytematic medical or nursing validation to confirm chemotherapy administration).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- front phase (Other): The current circuit remains unchanged (medical or nursing validation to confirm chemotherapy administration). Patient satisfaction is collected at each visit to the day hospital unit for chemotherapy.
  Interventions: Other: Standard follow up
- Post Phase (Other): A short circuit is set up. If no contraindications are identified by the plateform with the remote PRO collection, patients will undergo chemotherapy directly the next day (without any medical validation). Patient satisfaction is also collected at each visit to the day hospital unit for chemotherapy.
  Interventions: Other: short circuit

INTERVENTIONS:
Other: Standard follow up — Patients enrolled into front phase will be followed in a standard way without any additional procedure except satisfaction questionnaire
  Arms: front phase
Other: short circuit — Patients included in the post phase will have to complete the "cem@santé" application. If no contraindications are identified by the plateform with the remote PRO collection, patients will undergo chemotherapy directly the next day (without any medical validation).
  Arms: Post Phase

SUMMARY:
The present study proposes a new organization of the Day Hospital unit with several possible pathways defined by PRO.

The organization realies on a platform composed of nurses supervised by an IPA and a doctor one day before a treatment in the day hospitalization unit admission, results of PROs collectyed through the CEM@santé application (a French health care application) are reviewed by nurses from the platform and chemotherapy delivery is confirmed.

The study is planed in 2 steps.

1. st stage: the current circuit remains unchanged (with systematic medical or nursing validation to confirm chemotherapy administration. Patient satisfaction is collected at each visit to the day hospital unit for chemotherapy. 73 patients will be included in this phase.
2. nd stage: a short circuit is set up. If no contraindications are identified by the plateform with the remote PRO collection, patients will undergo chemotherapy directly the next day (without any medical validation. Patient satisfaction is also collected at each visit to the day hospital unit for chemotherapy. 73 patients will be included in this phase.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Patient treated for solid malignancy
* Patient starting a new chemotherapy or immunotherapy protocol.
* Patient receiving one of the following intravenous antineoplastic treatments in day hospital: Nivolumab(1), Pembrolizumab(1), Folfox(2), Folfirinox(2), Xelox Carboplatin, EC chemotherapy (Epirubicin/Cyclophosphamide)
* Affiliated and beneficiary to a social security system
* Informed and written consent

Note1: may be used in combination with tyrosine kinase inhibitors (TKIs) Note 2 :may be used in combination with bevacizumab, cetuximab or panitumumab

Exclusion Criteria:

* Patient treated in neo-adjuvant situation for breast cancer
* Does not have a connected device (smartphone, tablet or computer)
* Does not have an internet connection
* Difficulty in filling out a questionnaire
* Protected adult or deprived of her liberty
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Duration of stay in day hospital unit | Immediately after the chemotherapy
  Assess the impact on the duration of stay of an anticipated personalization of the stay in HDJ based on a platform of analysis of the PROs collected the day before and the implementation of a short circuit

SECONDARY OUTCOMES:
patient satisfaction | Immediately after the chemotherapy
  Assessed by EORTC OUT-PATSAT7 ( patient satisfaction with cancer care core questionnaire).
  satisfaction score between 0 (no satisfaction) and 100 (high satisfaction)
Caregiver satisfaction | Month3;Month6
  Assessed by self questionnaire
Health related patient quality of life | Immediately after the chemotherapy
  Assessed by EQ5D-5L (EuroQuol Five Dimension - Five Level Health Survey questionnaire) The scale has five subcomponents with scores from 1 (best) to 5 (worst)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de lutte contre le cancer Eugène Marquis, Rennes, France